CLINICAL TRIAL: NCT05348252
Title: Patient Journey Application for Discontinuing Inappropriate PPI Use: a Randomized Controlled Trial
Acronym: SUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N21.079
Record Dates: First submitted 2022-04-05; First posted 2022-04-27 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2022-04

CONDITIONS: Proton Pump Inhibitor; Inappropriate Drug Use; Discontinuation; E-health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Patient Journey App) (Experimental): The interventional group will receive all information and instructions on discontinuing PPI use through the Patient Journey App.
  Interventions: Other: Patient Journey App
- Control group (Conventional Care) (Active Comparator): The control group will receive all information and instructions on discontinuing PPI use through email as a digital information folder.
  Interventions: Other: Information folder

INTERVENTIONS:
Other: Patient Journey App — The group will receive all information and insctructions on discontinuing PPI use through the Patient Journey App which timely deliveres all information.
  Arms: Interventional group (Patient Journey App)
Other: Information folder — The group will receive all information and instructions on discontinuing PPI use through an information folder.
  Arms: Control group (Conventional Care)

SUMMARY:
Rationale/objective: This study hypothesizes that offering patient-tailored and dosed information on PPI discontinuation in patients with inappropriate chronic PPI use will result in an increased discontinuation rate when compared to a conventional information folder offering all information on discontinuing inappropriate PPI use at once.

Study design: Multicenter randomized controlled trial.

Study population: A minimum 152 patients with chronic PPI use without a valid indication for chronic PPI use according to the NHG-guidelines will be included. Possible participants will be identified at the outpatient clinics of the departments of Internal Medicine, Gastroenterology, Rheumatology and Nephrology in the Radboud University Medical Center, Canisius Wilhelmina Hospital and Sint Maartenskliniek.

Intervention: Timely informing patients on discontinuing PPI use through the Patient Journey App.

Control: Conventional information, consisting of an online information folder on discontinuing PPI use.

Inclusion criteria:

* Patients with daily PPI use for at least 4 weeks;
* Age 18-70 years.

Exclusion criteria:

* Chronic PPI indication according to NHG-guidelines;
* Chronic PPI indication according to treating physician, despite absence of chronic PPI indication according to NHG-guidelines;
* Patients that underwent anti-reflux surgery;
* No understanding of the study or study procedures including the digital application (smartphone/computer skills);
* No smartphone/computer available;
* No informed consent;
* Limited life span.

Primary end point:

- Discontinuation of PPI use at 2-month follow-up, defined as self-declared intake of a maximum of 1 tablet in the previous 14 days.

Secondary end points:

* Upper gastrointestinal symptoms or disorders that are potentially related to discontinuation of PPI use, subdivided as:

  * Upper gastrointestinal symptoms as measured by the Patient Assessment of Gastrointestinal Symptom Severity Score (PAGI-SYM);
  * Any upper gastrointestinal event that requires a doctor's visit or hospitalization.
* Potential adverse drug reactions (ADRs) of PPIs, subdivided as:

  * Most prevalent (1-10%) ADRs according to the Medicines Evaluation Board1: obstipation, diarrhea, meteorism, abdominal pain, nausea/vomitus, headache;
  * Other potential ADRs requiring a doctor's visit or hospitalization. The following disorders are considered as potentially related to PPI use: any pneumonia, gastroenteritis, vitamin B12 deficiency, iron deficiency, calcium deficiency, fractures, acute interstitial nephritis or hypomagnesaemia.
* Frequency of PPI use, measured monthly during follow-up, measured as number of PPI tablets per month;
* Start of new medication for upper gastrointestinal symptoms, other than PPI (e.g., antacids, H2-blockers, analgesics, anti-emetics);
* Association between successful discontinuation and variables such as gender, age, fear of ADRs, occurrence of potential ADRs or occurrence of rebound effect;
* Change in lifestyle (BMI, smoking status and alcohol usage);
* Patient Journey App usability as measured by the System Usability Score (SUS);
* Self-management behavior as measured by the short Patient Activation Measure (PAM-13);
* Recurrent PPI use, defined as the intake of more than 1 PPI tablet in the previous 14 days measured as self-declared intake during follow-up after successful discontinuation during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with daily PPI use for at least 4 weeks;
* Age 18-70 years.

Exclusion Criteria:

* Chronic PPI indication according to NHG-guidelines;
* Chronic PPI indication according to treating physician, despite absence of chronic PPI indication according to NHG-guidelines;
* Patients that underwent anti-reflux surgery;
* No understanding of the study or study procedures including the digital application (smartphone/computer skills);
* No smartphone/computer available;
* No informed consent;
* Limited life span.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Discontinuation rate | At 2 months follow-up
  Succesful discontinuation of PPI use

SECONDARY OUTCOMES:
Upper gastrointestinal symptoms | 2 monthly up to 12 months
  Change in upper gastrointestinal symptoms or disorders that are potentially related to discontinuation of PPI use
Adverse drug reactions | 2 monthly up to 12 months
  Change in potential adverse drug reactions (ADRs) of PPIs
Frequency of PPI use | Monthly up to 12 months
  Change in frequency of PPI use
New medication | Monthly up to 12 months
  Start of new medication for upper gastrointestinal symptoms, other than PPI (e.g., antacids, H2-blockers, analgesics, anti-emetics)
Association betwee succesful discontinuation of PPIs and patient characteristics | At 2 months follow-up
  Association between successful discontinuation and variables such as gender, age, fear of ADRs, occurrence of potential ADRs or occurrence of rebound effect. Fear of ADRs will be evaluated at baseline as a yes/no question. Occurrence of potential ADRs will be measured at 2 months follow-up by asking if patients experience adverse drug reactions that have been registered in 1-10% of users. Occurrence of rebound effect will be measured according to the PAGI-SYM questionnaire.
Lifestyle change | 2 monthly up to 12 months
  Change in lifestyle (BMI, smoking status and alcohol usage)
App usability | At 4 months follow-up
  Patient Journey App usability as measured by the System Usability Score (SUS)
Self-management behavior | 2 monthly up to 12 months
  Change in self-management behavior as measured by the short Patient Activation Measure (PAM-13)
Recurrent PPI use | Monthly up to 12 months
  Recurrent PPI use

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes